CLINICAL TRIAL: NCT00609908
Title: The Technique of Skin Stretching for Acute Burn Treatment and Scar Reconstruction: Clinical Applications and Working Mechanisms.
Brief Title: The Technique of Skin Stretching for Acute Burn Treatment and Scar Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Responsible Party: Association of Dutch Burn Centres, Association of Dutch Burn Centres
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06.201; 06.201
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Burns; Scars
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (Active Comparator): Acute Burn Wounds: Wound debridement and split skin grafting
  Interventions: Procedure: Split skin graft
- A2 (Experimental): Acute Burn Wounds: excision of the burn wound and primary closure, using a skin stretching device
  Interventions: Procedure: skin stretching device
- B1 (Active Comparator): Scar reconstruction: serial excision
  Interventions: Procedure: serial excision
- B2 (Experimental): Scar reconstruction: primary closure, using skin stretching device
  Interventions: Procedure: skin stretching device

INTERVENTIONS:
Procedure: Split skin graft — After wound bed preparation the skin defect is covered with a skin transplant (split skin graft)
  Arms: A1
Procedure: skin stretching device — after woundbed preparation the wound is primarily closed by aid of the skin stretching device
  Arms: A2
Procedure: serial excision — as much scar as possible is excised, whereafter the wound is closed
  Arms: B1
Procedure: skin stretching device — after the scar is excised, the wound is primarily closed by aid of the skin stretching device
  Arms: B2

SUMMARY:
Objective:

A randomized controlled trial is performed to evaluate the clinical effectiveness of the skin stretching technique for two categories:

1. acute burn wounds: wound closure by means of skin stretching should lead to a significant reduction of scar surface area in comparison to the standard technique, the split skin grafting;
2. scar reconstructions: wound closure by means of skin stretching during one operative procedure should lead to a comparable scar surface in comparison to the multiple procedures techniques such as serial excision.

Study design:

Skin stretching will be compared to split skin grafting and should result in burn wound closure with significantly smaller scars. Also, a comparison will be made between the technique of serial excision versus skin stretching for scar reconstructions.

Scar evaluation three and twelve months after surgery will include the following parameters:

* surface area;
* Patient and Observer Scar Assessment Scale (POSAS);
* elasticity;
* vascularization and pigmentation;
* thickness;
* dermal architecture.

After 12 months adults will undergo a biopsy of the scar under local anesthesia. The experimental group, treated with the skin stretcher will undergo one extra biopsy of the formerly stretched skin.

Intervention:

At the start of the operation will be determined by randomization if skin stretching or split skin grafting (acute burn wounds) or serial excision (scar reconstruction category) will be performed.

DETAILED DESCRIPTION:
Eligibility criteria:

Inclusion:

1. Acute Burn wounds or scar reconstructions that require surgical treatment; 2. Sufficient healthy skin at (at least) one edge of the wound/scar must be available for the stretching procedure.

3. Age >= 18 years

Exclusion:

1. language barrier;
2. known history of keloid formation;
3. systemic diseases: Diabetes Mellitus, immunodeficiency, arterial insufficiency;
4. local or systemic application of corticosteroids;
5. psychiatric diseases leading to study bias (e.g. automutilation);
6. skin diseases that lead to collagen and/or elastin abnormalities such as Ehlers Danlos;
7. radiated skin;
8. wound located at extremities, exceeding >33% of circumference (acute burn category);

Primary study parameters/outcome of the study:

The primary study parameter is the surface area of the scar after 12 months

Secondary study parameters/outcome of the study (if applicable):

All scars will also be subjected to the scar evaluation protocol after 3 and 12 months by an independent observer for the evaluation of the:

* patient and observer scar assessment scale (POSAS);
* scar elasticity (Cutometer);
* scar vascularisation & pigmentation (DermaSpectrometer);
* scar thickness (histopathology, only after 12 months).

Punch biopsies are taken for morphometry of dermal architecture (Fourier analysis). During surgery one biopsy is obtained of the normal skin. In the experimental group an additional biopsy is obtained at the end of the stretching procedure in order to be able to compare structure of the dermal matrix and orientation of the collagen fibers.

After 1 year, one biopsy is taken from the scar. The experimental group will undergo one additional biopsy of the formerly stretched skin.

ELIGIBILITY:
Inclusion criteria:

* Acute Burn wounds or scar reconstructions that require surgical treatment;
* Sufficient healthy skin at (at least) one edge of the wound/scar must be available for the stretching procedure;
* Age >= 18 years.

Exclusion criteria:

* Language barrier;
* Known history of keloid formation;
* Systemic diseases: Diabetes Mellitus, immunodeficiency, arterial insufficiency;
* Local or systemic application of corticosteroids;
* Psychiatric diseases leading to study bias (e.g. automutilation);
* Skin diseases that lead to collagen and/or elastin abnormalities such as Ehlers Danlos;
* Radiated skin;
* Wound located at extremities, exceeding >33% of circumference (acute burn category).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the surface area of the scar after 12 months | 3 and 12 months after surgery

SECONDARY OUTCOMES:
scar evaluation protocol: - patient and observer scar assessment scale (POSAS); - scar elasticity (Cutometer); - scar vascularization & pigmentation (DermaSpectrometer); - scar thickness | 3 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: E Middelkoop, Professor, Principal Investigator — VU MC; P.P.M. van Zuijlen, MD, PhD, Study Director — Red Cross Hospital Beverwijk
Locations (1):
- Red Cross Hospital, Beverwijk, Netherlands